CLINICAL TRIAL: NCT01833793
Title: Mirena and Amenorrhea Related acceptabILity in Contraception indIcAtion
Brief Title: Descriptive, Prospective, Non-interventional Study (NIS) to Describe Mirena and Amenorrhea Related Acceptability in Contraception Indication in Medical Practice
Acronym: MARILIA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16314; MA1211DZ (Other: Company internal)
Record Dates: First submitted 2013-03-13; First posted 2013-04-17 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Female Contraception
Keywords: Mirena; Contraception; Amenorrhea
MeSH Terms: conditions — Amenorrhea | interventions — Levonorgestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Levonorgestrel IUD (Mirena, BAY86-5028)

INTERVENTIONS:
Drug: Levonorgestrel IUD (Mirena, BAY86-5028) — Women who have been prescribed Mirena in contraception; followed up for 12 months

SUMMARY:
MARILIA is a prospective, non-interventional, multicenter study. The purpose of this study is to describe the acceptability of Amenorrhea in contraception indication of Mirena users during one year follow up in medical practice. 500 patients in 20 centers will be enrolled in the study. Bleeding profile, removal or non-removal of the IUS (IntraUterine System) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-40 years at the time of Mirena IUD insertion
* Using Mirena only for contraception indication
* Never having used the product before
* No heavy menstrual bleeding diagnosed
* Have signed informed consent to participate in this study

Exclusion Criteria:

* Nulliparous
* Pregnancy
* Mirena's contre-indication
* Mirena for HMB
* Abnormal bleeding pattern

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women who have been prescribed Mirena for contraception.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-02; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Proportion of Mirena users who have at least one period of Amenorrhea of at least three months | 12 months
Cumulative incidence rate of Amenorrhea over the duration of follow up period in Mirena users | 12 months

SECONDARY OUTCOMES:
Proportion of Mirena users who have menstrual disorders | 12 months
Proportion of Mirena users with menorrhagia | 12 months
Cumulative rate of satisfaction in Mirena users | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Algeria